CLINICAL TRIAL: NCT06372925
Title: A Multi-Center, Randomized, Open-label, Parallel, Controlled Phase Ⅳ Clinical Trial to Evaluate the Effect of Inclisiran on Coronary Atherosclerotic Plaque in Patients With Acute Myocardial Infarction and Elevated Low-density Lipoprotein Cholesterol
Brief Title: Intravascular Imaging Study of the Effect of Inclisiran on Plaque in Patients With Acute Myocardial Infarction
Acronym: V-ACCELERATE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKJX839A1CN04; CKJX839A1CN04 (Other: Novartis)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Plaque, Atherosclerotic
Keywords: Acute myocardial infarction,; Atherosclerotic plaque,; Inclisiran,; IVUS,; OCT,; PCI
MeSH Terms: conditions — Plaque, Atherosclerotic | interventions — Atorvastatin; ALN-PCS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: IVUS/OCT will be conducted in local lab and blinded analyzed to Independent Review Committee(IRC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclisiran and atorvastatin (Experimental): Inclisiran 284mg SC (at D1,D90,D270)+ 20mg atorvastatin PO
  Interventions: Drug: atorvastatin; Procedure: IVUS/OCT; Drug: inclisiran
- atorvastatin (Active Comparator): 20mg atorvastatin PO
  Interventions: Drug: atorvastatin; Procedure: IVUS/OCT

INTERVENTIONS:
Drug: atorvastatin — 20mg atorvastatin PO
Procedure: IVUS/OCT — performed the IVUS/OCT at baseline and Day 360
Drug: inclisiran — Inclisiran 284mg SC
  Arms: Inclisiran and atorvastatin

SUMMARY:
This study is to evaluate the effect of Inclisiran on coronary atherosclerosis using intravascular ultrasound (IVUS) and optical coherence tomography (OCT) in patients with acute myocardial infarction and elevated low-density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
This study will be a multi-center, randomized, parallel-group, open-label, phase 4 study. Participants will be approximately 318 Chinese adults diagnosed with new-onset STEMI/NSTEMI and elevated LDL-C (LDL-C > 1.8 mmol/L if on stable dose of statin (with or without ezetimibe) for ≥ 4 weeks; LDL-C > 2.6 mmol/L if not on stable dose of statin (with or without ezetimibe) for ≥ 4 weeks). Participants will be 1:1 randomized to investigational group (Inclisiran 284mg + 20mg atorvastatin) or control group (20mg atorvastatin) for 360 days. Participants and investigator will be unblinded to the identity of the treatment from the time of randomization. Independent Review Committee (IRC) staff performing the study assessments (IVUS and OCT analysis) will be blinded to the identity of the treatment from the time of randomization until final database lock.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 and ≤ 75 years of age.
2. Acute myocardial infarction (STEMI ≤ 24h/NSTEMI ≤ 72h of onset of symptoms) with planned PCI.
3. At least 1 major, non-infarct-related coronary artery ("target vessel") meet all of the following criteria judged by the investigator:

1) Presence of atherosclerotic plaque with ≥ 20% and ≤ 50% diameter stenosis by coronary angiography.

2) Target vessel deemed to be accessible to imaging catheters and suitable for intravascular imaging in the proximal (50 mm) segment ("target segment") 3) Target vessel is suitable for IVUS and OCT evaluation. 4) Not have undergone previous PCI within target vessel. 5) Not be a bypass graft or a bypassed native vessel. 4. Rapid LDL-C test value at screening period of:

1. LDL-C > 1.8 mmol/L if on stable dose of statin (with or without ezetimibe) for ≥ 4 weeks upon signing ICF.
2. LDL-C > 2.6 mmol/L if not on stable dose of statin (with or without ezetimibe) for ≥ 4 weeks upon signing ICF.

5. Written informed consent must be obtained.

Exclusion Criteria:

1. Familial hypercholesterolemia or secondary hypercholesterolemia.
2. Clinically instable AMI (hemodynamic or electrical instability).
3. Left main disease, defined as ≥ 50% diameter stenosis of the left main coronary artery by coronary angiography.
4. Three-vessel disease, defined as ≥ 70% diameter stenosis of 3 major epicardial coronary vessels or in major branches of these arteries by coronary angiography.
5. Have a plan for interventional procedure within 12 months after signing ICF.
6. Known intolerance to Atorvastatin OR known statin intolerance.
7. Patients already on high-intensity statin including atorvastatin 40 or 80 mg or rosuvastatin 20 mg upon signing ICF.
8. Patients not suitable for IVUS/OCT evaluation (e.g., significant calcification , etc) judged by the investigator.
9. Patients qualify for coronary artery bypass surgery at screening and history of coronary artery bypass surgery.
10. Cardiac disorders:

1) Uncontrolled cardiac arrhythmia, defined as recurrent and symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response not controlled by medications in the past 3 months prior to screening; 2) Pacemaker or ICD in situ; and/or 3) Uncontrolled severe hypertension with systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to randomization despite antihypertensive therapy.

11. Rapid lipid test triglyceride (TG) level > 400mg/dL (4.5 mmol/L) at screening.

12. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in alanine aminotransferase (ALT), aspartate aminotransferase (AST), > 3x the upper limit of normal (ULN), or total bilirubin > 2x ULN before the randomization.

13. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2(Calculated according to the modified MDRD equation).

14. Severe concomitant non-cardiovascular disease that carries the risk of reducing life expectancy to less than 2 years.

15. Previous (within 90 days before randomization), current or planned treatment with a PCSK9 monoclonal antibody (mAb).

16. Previous exposure to Inclisiran or any other non-mAb PCSK9-targeted therapy 2 years prior to randomization.

17. Participation in another investigational device or drug study currently, or within 5 half-live (if drug) or 30 days whichever is longer, prior to randomization.

18. History of hypersensitivity to any study drug or its excipients. 19. Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study and/or put the participant at significant risk according to investigator's judgment.

20. Pregnant or nursing (lactating) women. 21. Women of child-bearing potential, unless they are using effective methods of contraception during study treatment.

22. Any conditions that according to the investigator could interfere with the conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Change in percent atheroma volume (PAV) | Up to 360 days
  Change in PAV assessed by intravascular ultrasound (IVUS) from baseline to Day 360.

SECONDARY OUTCOMES:
Change in minimum fibrous cap thickness (FCT) | Up to 360 days
  Change in minimum FCT as determined by optical coherence tomography (OCT) from baseline to Day 360
Change in mean minimum FCT of all images | 360 days
  Change in mean minimum fibrous cap thickness (FCT) of all images as determined by OCT from baseline to Day 360.
Change in normalized total atheroma volume (NTAV) | Up to 360 days
  Change in NTAV as determined by intravascular ultrasound (IVUS) from baseline to Day 360
Proportion of participants with progression, regression, or no change in PAV | Up to 360 days
  Proportion of participants with progression, regression, or no change in percent atheroma volume (PAV) at Day 360
Change in LDL-C | Baseline, Day 30, Day 150 and Day 360
  Change in low-density lipoprotein cholesterol (LDL-C)
Change in TC | Baseline, Day 30, Day 150 and Day 360
  Change in total cholesterol (TC).
Change in HDL-C | Baseline, Day 30, Day 150 and Day 360
  Change in high-density lipoprotein cholesterol (HDL-C).
Change in non-HDL-C | Baseline, Day 30, Day 150 and Day 360
  Change in non-high-density lipoprotein cholesterol (non-HDL-C).
Change in ApoB | Baseline, Day 30, Day 150 and Day 360
  Change in apolipoprotein B (ApoB).
Change in ApoA1 | Baseline, Day 30, Day 150 and Day 360
  Change in apolipoprotein A1 (ApoA1).
Change in Lp(a) | Baseline, Day 30, Day 150 and Day 360
  Change in lipoprotein (a) (Lp(a))
Change in TG | Baseline, Day 30, Day 150 and Day 360
  Change in triglycerides (TG)
Proportion of participants with LDL-C target attainment | Day 30, Day 150 and Day 360
  Proportion of participants with LDL-C target attainment at Day 30, Day 150, and Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- China (18):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Zunyi, Guizhou
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Jining, Shandong
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Lanzhou
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com